CLINICAL TRIAL: NCT03829332
Title: A Phase 3, Randomized, Double-blind Trial of Pembrolizumab (MK-3475) With or Without Lenvatinib (E7080/MK-7902) in Participants With Treatment-naïve, Metastatic Nonsmall Cell Lung Cancer (NSCLC) Whose Tumors Have a Tumor Proportion Score (TPS) Greater Than or Equal to 1% (LEAP-007)
Brief Title: Efficacy and Safety Study of Pembrolizumab (MK-3475) With or Without Lenvatinib (MK-7902/E7080) in Adults With Programmed Cell Death-Ligand 1 (PD-L1)-Positive Treatment-naïve Nonsmall Cell Lung Cancer (NSCLC) (MK-7902-007/E7080-G000-314/LEAP-007)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7902-007; MK-7902-007 (Other: MSD); E7080-G000-314 (Other: Eisai Protocol Number); LEAP-007 (Other: MSD); 194670 (Registry Identifier: JAPIC-CTI); 2018-003794-98 (EudraCT Number)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death-ligand 1 (PD-L1, PDL1); programmed cell death-ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Lenvatinib (Experimental): Participants receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily (QD) on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- Pembrolizumab + Placebo (Active Comparator): Participants receive pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule QD on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Placebo for lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Lenvatinib — oral capsule
  Other Names: MK-7902; E7080; LENVIMA®
  Arms: Pembrolizumab + Lenvatinib
Drug: Placebo for lenvatinib — oral capsule
  Arms: Pembrolizumab + Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of pembrolizumab (MK-3475) combined with lenvatinib (MK-7902/E7080) compared to pembrolizumab alone (with placebo for lenvatinib) in treatment-naïve adults with no prior systemic therapy for their metastatic non-small cell lung cancer (NSCLC) whose tumors have a programmed cell death-ligand 1 (PD-L1) Tumor Proportion Score (TPS) greater than or equal to 1%.

The primary study hypotheses are that: 1) the combination of pembrolizumab and lenvatinib is superior to pembrolizumab alone as assessed by Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1); and 2) the combination of pembrolizumab and lenvatinib is superior to pembrolizumab alone as assessed by Overall Survival (OS).

DETAILED DESCRIPTION:
As of 30-Jul-2021, active participants, investigator, and sponsor personnel or delegate(s) involved in the treatment administration or clinical evaluation of the participants will be unblinded. Participants will discontinue lenvatinib and placebo, and participants who remain on treatment will receive open-label pembrolizumab only.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC)
* Has Stage IV NSCLC (American Joint Committee on Cancer [AJCC 8th edition])
* Has measurable disease based on RECIST 1.1
* Has tumor tissue that demonstrates programmed cell death-ligand 1 (PD-L1) expression in ≥1% of tumor cells (Tumor Proportion Score [TPS] ≥1%) as assessed by immunohistochemistry (IHC) 22C3 pharmDx assay (Dako North America, Inc.) at a central laboratory
* Has a life expectancy of ≥3 months
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days before the first dose of study treatment but before randomization
* Male participants must agree to the following during the treatment period and for ≥7 days after the last dose of lenvatinib/matching placebo: 1) Be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent, OR 2) Must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause)
* Female participants are eligible to participate if not pregnant or breastfeeding, and ≥1 of the following applies: 1) Is not a woman of child-bearing potential (WOCBP), OR 2) Is a WOCBP and is using a highly effective contraceptive method that has a low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle during the treatment period and for ≥120 days post pembrolizumab or ≥30 days post lenvatinib/matching placebo, whichever occurs last
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mm Hg and no change in antihypertensive medications within 1 week before randomization
* Has adequate organ function

Exclusion Criteria:

* Has known untreated central nervous system metastases and/or carcinomatous meningitis
* Has active hemoptysis (at least 0.5 teaspoon of bright red blood) within 2 weeks prior to the first dose of study intervention
* Has radiographic evidence of intratumoral cavitations, encasement, or invasion of a major blood vessel
* Has a known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for ≥3 years since initiation of that therapy. (Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.)
* Has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Has had an allogeneic tissue/solid organ transplant
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a history of (noninfectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease
* Has a known history of hepatitis B or known active hepatitis C virus infection
* Has a history of a gastrointestinal condition or procedure that in the opinion of the investigator may affect oral study drug absorption.
* Has significant cardiovascular impairment within 12 months of the first dose of study treatment, such as a history of congestive heart failure greater than New York Heart Association Class II, unstable angina, myocardial infarction, cerebrovascular accident/stroke, or cardiac arrhythmia associated with hemodynamic instability
* Has not recovered adequately from any toxicity and/or complications from major surgery before starting study treatment
* Has a known history of active tuberculosis (TB)
* Has an active infection requiring systemic therapy
* Has previously had a severe hypersensitivity reaction to treatment with a monoclonal antibody or has a known sensitivity or intolerance to any component of lenvatinib or pembrolizumab
* Has received prior systemic chemotherapy or other targeted or biological antineoplastic therapy for their metastatic NSCLC
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], Tumor necrosis factor receptor superfamily, member 4 [OX 40], tumor necrosis factor receptor superfamily member 9 [CD137]) or has received lenvatinib as monotherapy or in combination with anti- programmed cell death protein (anti-PD-1) agents
* Has received radiotherapy within 14 days before the first dose of study treatment or received lung radiation therapy of >30 Gray (Gy) within 6 months before the first dose of study treatment. (Note: Participants must have recovered from all radiation-related toxicities to ≤Grade 1, not require corticosteroids, and not have had radiation pneumonitis.)
* Has a diagnosis of immunodeficiency or is receiving any form of immunosuppressive therapy within 7 days before the first dose of study treatment
* Is receiving systemic steroid therapy (doses >10 mg daily of prednisone equivalent) within 7 days before the first dose of study treatment
* Has received a live or attenuated vaccine within 30 days before the first dose of study treatment
* Has had major surgery within 3 weeks prior to first dose of study treatment
* Has pre-existing ≥Grade 3 gastrointestinal or nongastrointestinal fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (162):
- United States (18):
  - Alaska Clinical Research Center ( Site 0511), Anchorage, Alaska
  - Ironwood Cancer & Research Centers ( Site 0541), Chandler, Arizona
  - CBCC Global Research, Inc. ( Site 0532), Bakersfield, California
  - Scripps Cancer Center ( Site 0521), La Jolla, California
  - Florida Hospital ( Site 0526), Orlando, Florida
  - Northwest Georgia Oncology Centers PC ( Site 0518), Marietta, Georgia
  - Illinois Cancer Care, PC ( Site 0557), Peoria, Illinois
  - Parkview Cancer Center ( Site 0542), Fort Wayne, Indiana
  - University of Kentucky School of Medicine & Hospitals ( Site 0517), Lexington, Kentucky
  - Anne Arundel Medical Center Oncology and Hematology ( Site 0514), Annapolis, Maryland
  - Munson Medical Center ( Site 0512), Traverse City, Michigan
  - Park Nicollet Frauenshuh Cancer Center ( Site 0554), Saint Louis Park, Minnesota
  - University of Missouri Health Care ( Site 0555), Columbia, Missouri
  - Billings Clinic Cancer Center ( Site 0508), Billings, Montana
  - Cone Health Cancer Center at Alamance Regional ( Site 0527), Greensboro, North Carolina
  - Genesis Cancer Care Center ( Site 0559), Zanesville, Ohio
  - Oregon Health Sciences University ( Site 0544), Portland, Oregon
  - Central Texas Veterans Healthcare System ( Site 0533), Temple, Texas
- Australia (5):
  - Orange Health Services ( Site 0002), Orange, New South Wales
  - Wollongong Private Hospital ( Site 0005), Wollongong, New South Wales
  - The Prince Charles Hospital ( Site 0011), Chermside, Queensland
  - Ballarat Oncology and Haematology Services ( Site 0008), Wendouree, Victoria
  - St John of God Murdoch Medical Clinic ( Site 0001), Perth, Western Australia
- Canada (5):
  - Cross Cancer Institute ( Site 0400), Edmonton, Alberta
  - Lions Gate Hospital ( Site 0407), North Vancouver, British Columbia
  - William Osler Health System (Brampton Civic Hospital) ( Site 0402), Brampton, Ontario
  - Windsor Regional Cancer Program ( Site 0404), Windsor, Ontario
  - McGill University Health Centre ( Site 0418), Montreal, Quebec
- China (17):
  - Beijing Chest Hospital Capital Medical University ( Site 0111), Beijing, Anhui
  - Anhui Provincial Hospital ( Site 0108), Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University ( Site 0113), Hefei, Anhui
  - Peking Union Medical College Hospital ( Site 0105), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0102), Beijing, Beijing Municipality
  - Xiangya Hospital of Central South University ( Site 0115), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0104), Changsha, Hunan
  - Jiangsu Cancer Hospital ( Site 0101), Nanjing, Jiangsu
  - The First Hospital of Jilin University ( Site 0110), Changchun, Jilin
  - Zhongshan Hospital Fudan University ( Site 0100), Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital ( Site 0112), Shanghai, Shanghai Municipality
  - 1st Affil Hosp of Med College of Xi'an Jiaotong University ( Site 0103), XiAn, Shanxi
  - West China Hospital of Sichuan University ( Site 0117), Chengdu, Sichuan
  - The First Affiliated Hospital Zhejiang University ( Site 0106), Hangzhou, Zhejiang
  - Hangzhou First People's Hospital ( Site 0109), Hangzhou, Zhejiang
  - 2nd Affil Hosp of Zhejiang University College of Medicine ( Site 0114), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0116), Hangzhou, Zhejiang
- Colombia (6):
  - Hospital General de Medellin Luz Castro de Gutierrez ( Site 0368), Medellín, Antioquia
  - Fundacion Centro de Investigacion Clinica CIC ( Site 0366), Medellín, Antioquia
  - Biomelab S A S ( Site 0365), Barranquilla, Atlántico
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 0374), Valledupar, Cesar Department
  - Oncomedica S.A. ( Site 0372), Montería, Departamento de Córdoba
  - Centro Medico Imbanaco de Cali S.A ( Site 0369), Cali, Valle del Cauca Department
- Estonia (3):
  - AS Ida-Tallinna Keskhaigla ( Site 0161), Tallinn, Harju
  - SA Pohja-Eesti Regionaalhaigla ( Site 0162), Tallinn, Harju
  - SA Tartu Ulikooli Kliinikum ( Site 0160), Tartu, Tartu
- France (10):
  - CHU Jean Minjoz ( Site 0167), Besançon, Doubs
  - Institut Curie - Centre Rene Huguenin ( Site 0181), Saint-Cloud, Hauts-de-Seine
  - ICM Val D Auerelle ( Site 0177), Montpellier, Herault
  - CHU de Grenoble - Hopital Michallon ( Site 0169), La Tronche, Isere
  - Institut de Cancerologie de l Ouest Centre Rene Gauducheau ( Site 0185), Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier de la Cote Basque ( Site 0173), Bayonne, Pyrenees-Atlantiques
  - CHU de Rouen ( Site 0174), Rouen, Seine-Maritime
  - CHU Amiens Sud ( Site 0182), Amiens, Somme
  - Centre hospitalier Toulon Sainte-Musse ( Site 0172), Toulon, Var
  - Institut Curie ( Site 0166), Paris
- Hungary (8):
  - Bekes Megyei Kozponti Korhaz - Pandy Kalman Tagkorhaza ( Site 0207), Gyula, Bekes County
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktatokorhaz ( Site 0202), Miskolc, Borsod-Abauj Zemplen county
  - CRU Hungary KFT ( Site 0209), Miskolc, Borsod-Abauj Zemplen county
  - Petz Aladar Megyei Oktato Korhaz ( Site 0213), Győr, Győr-Moson-Sopron
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 0203), Szolnok, Jász-Nagykun-Szolnok
  - Tudogyogyintezet Torokbalint ( Site 0205), Törökbálint, Pest County
  - Semmelweis Egyetem ( Site 0210), Budapest
  - Somogy Megyei Kaposi Mor Oktato Korhaz ( Site 0217), Kaposvár
- Israel (8):
  - Bnei Zion Medical Center ( Site 0227), Haifa, Heifa
  - Sheba Medical Center ( Site 0220), Ramat Gan, Tel Aviv
  - Soroka Medical Center ( Site 0222), Beersheba
  - Rambam Medical Center ( Site 0223), Haifa
  - Meir Medical Center ( Site 0221), Kfar Saba
  - Rabin Medical Center ( Site 0224), Petah Tikva
  - Sourasky Medical Center ( Site 0225), Tel Aviv
  - Barzilai Medical Center ( Site 0226), Ashkelon, Ḥeifā
- Italy (8):
  - Azienda Ospedaliera S. Giovanni Addolorata-Oncologia Medica ( Site 0233), Rome, Lazio
  - Presidio Ospedaliero San Vincenzo ( Site 0231), Taormina, Messina
  - Centro di Riferimento Oncologico CRO ( Site 0235), Aviano, Pordenone
  - Azienda Ospedaliera San Giuseppe Moscati ( Site 0234), Avellino
  - Universita Magna Grecia ( Site 0230), Catanzaro
  - A.O. Universitaria Careggi ( Site 0236), Florence
  - Ospedale Santa Maria delle Croci ( Site 0232), Ravenna
  - Policlinico Gemelli di Roma ( Site 0237), Roma
- Japan (16):
  - Aichi Cancer Center Hospital ( Site 0018), Nagoya, Aichi-ken
  - Kurume University Hospital ( Site 0025), Kurume, Fukuoka
  - Hyogo Cancer Center ( Site 0021), Akashi, Hyōgo
  - Kanagawa Cardiovascular and Respiratory Center ( Site 0026), Yokohama, Kanagawa
  - Kanagawa Cancer Center ( Site 0023), Yokohama, Kanagawa
  - Miyagi Cancer Center ( Site 0028), Natori-shi, Miyagi
  - Sendai Kousei Hospital ( Site 0022), Sendai, Miyagi
  - National Hospital Organization Kinki-chuo Chest Medical Center ( Site 0027), Sakai, Osaka
  - Kindai University Hospital ( Site 0017), Sayama, Osaka
  - National Hospital Organization Kyushu Medical Center ( Site 0015), Fukuoka
  - Kyushu University Hospital ( Site 0030), Fukuoka
  - Okayama University Hospital ( Site 0020), Okayama
  - Osaka International Cancer Institute ( Site 0019), Osaka
  - Toranomon Hospital ( Site 0016), Tokyo
  - Juntendo University Hospital ( Site 0029), Tokyo
  - Nippon Medical School Hospital ( Site 0024), Tokyo
- Malaysia (7):
  - Hospital Tengku Ampuan Afzan ( Site 0062), Kuantan, Pahang
  - Hospital Pulau Pinang. ( Site 0065), George Town, Pulau Pinang
  - Institut Kanser Negara - National Cancer Institute ( Site 0063), Putrajaya, Putrajaya
  - Sarawak General Hospital ( Site 0064), Kuching, Sarawak
  - Beacon Hospital Sdn Bhd ( Site 0067), Petaling Jaya, Selangor
  - University Malaya Medical Centre ( Site 0061), Kuala Lumpur
  - Gleneagles Penang ( Site 0066), Pulau Pinang
- Mexico (5):
  - Consultorios de Medicina Especializada del Sector Privado ( Site 0388), Guadalajara, Jalisco
  - Medica Sur S.A.B de C.V. ( Site 0384), Mexico City, Mexico City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares ( Site 0381), Madero, Tamaulipas
  - Instituto Nacional de Cancerologia. ( Site 0382), Mexico City
  - Oaxaca Site Management Organization SC ( Site 0389), Oaxaca City
- Poland (8):
  - Ars Medical Sp. z o.o. ( Site 0254), Piła, Greater Poland Voivodeship
  - Krakowski Szpital Specjalistyczny im Jana Pawla II ( Site 0253), Krakow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie ( Site 0243), Krakow, Lesser Poland Voivodeship
  - Szpital Uniwersytecki im. Karola Marcinkowskiego ( Site 0247), Zielona Góra, Lubusz Voivodeship
  - Centrum Medyczne Pratia Ostroleka ( Site 0242), Ostrołęka, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 0252), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 0250), Przemyśl, Podkarpackie Voivodeship
  - SPZOZ USK nr 1 im. Norberta Barlickiego UM w Lodzi ( Site 0256), Lodz, Łódź Voivodeship
- Russia (7):
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 0262), Ufa, Baskortostan, Respublika
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 0266), Krasnoyarsk, Krasnoyarsk Krai
  - SBHI Samara Regional Clinical Oncology Dispensary ( Site 0265), Samara, Samara Oblast
  - SBHI Leningrad Regional Clinical Hospital ( Site 0263), Saint Petersburg, Sankt-Peterburg
  - Railway Hospital of OJSC ( Site 0268), Saint Petersburg, Sankt-Peterburg
  - City Clinical Oncology Center ( Site 0260), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 0269), Kazan', Tatarstan, Respublika
- South Korea (5):
  - Seoul National University Bundang Hospital ( Site 0075), Seongnam-si, Kyonggi-do
  - Chungbuk National University Hospital ( Site 0079), Cheongju-si, North Chungcheong
  - Ulsan University Hospital ( Site 0077), Ulsan, Ulsan-Kwangyokshi
  - Asan Medical Center ( Site 0076), Seoul
  - SMG-SNU Boramae Medical Center ( Site 0078), Seoul
- Taiwan (6):
  - National Taiwan University Hospital Hsin-Chu Branch ( Site 0087), Hsinchu
  - Taipei Medical University Shuang Ho Hospital ( Site 0090), New Taipei City
  - National Cheng Kung University Hospital ( Site 0086), Tainan
  - National Taiwan University Hospital ( Site 0088), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 0091), Taipei
  - Taipei Veterans General Hospital ( Site 0089), Taipei
- Turkey (Türkiye) (9):
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi ( Site 0321), Konya, Adana
  - Gulhane Egitim ve Arastirma Hastanesi ( Site 0316), Ankara
  - Abdurrahman Yurtaslan Onkoloji Hastanesi ( Site 0318), Ankara
  - Baskent Universitesi Ankara Hastanesi ( Site 0319), Ankara
  - Antalya Memorial Hospital Department of Medical Oncology ( Site 0324), Antalya
  - Akdeniz Universitesi Tip Fakultesi ( Site 0322), Antalya
  - Dokuz Eylul Universitesi Arastirma Uygulama Hastanesi ( Site 0314), Izmir
  - Sakarya Universitesi Egitim ve Arastirma Hastanesi ( Site 0323), Sakarya
  - Samsun Medical Park Hastanesi ( Site 0320), Samsun
- Ukraine (11):
  - Cherkasy Regional Hospital ( Site 0336), Cherkasy, Cherkasy Oblast
  - City Clinical Hosp.4 of DCC ( Site 0338), Dnipro, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 0346), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Regional Centre of Oncology-Thoracic organs ( Site 0337), Kharkiv, Kharkivs’ka Oblast’
  - Ukranian Center of TomoTherapy ( Site 0344), Kropyvnytskiy, Kirovohrad Oblast
  - Medical Center Verum ( Site 0334), Kyiv, Kyivska Oblast
  - Kyiv City Clinical Oncology Centre ( Site 0339), Kyiv, Kyivska Oblast
  - Medical and Diagnostic Centre LLC Dobryi Prognoz ( Site 0331), Kyiv, Kyivska Oblast
  - Lviv State Oncology Regional Treatment and Diagnostic Center ( Site 0341), Lviv, Lviv Oblast
  - MI Odessa Regional Oncological Centre ( Site 0333), Odesa, Odesa Oblast
  - Podillya Regional Center of Oncology ( Site 0343), Vinnytsia, Vinnytsia Oblast

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Yang JC, Han B, De La Mora Jimenez E, Lee JS, Koralewski P, Karadurmus N, Sugawara S, Livi L, Basappa NS, Quantin X, Dudnik J, Ortiz DM, Mekhail T, Okpara CE, Dutcus C, Zimmer Z, Samkari A, Bhagwati N, Csoszi T. Pembrolizumab With or Without Lenvatinib for First-Line Metastatic NSCLC With Programmed Cell Death-Ligand 1 Tumor Proportion Score of at least 1% (LEAP-007): A Randomized, Double-Blind, Phase 3 Trial. J Thorac Oncol. 2024 Jun;19(6):941-953. doi: 10.1016/j.jtho.2023.12.023. Epub 2023 Dec 29. PMID 38159809
- [Derived] Taylor MH, Schmidt EV, Dutcus C, Pinheiro EM, Funahashi Y, Lubiniecki G, Rasco D. The LEAP program: lenvatinib plus pembrolizumab for the treatment of advanced solid tumors. Future Oncol. 2021 Feb;17(6):637-648. doi: 10.2217/fon-2020-0937. Epub 2020 Dec 10. PMID 33300372
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 623 total participants randomized in the MK-7902-007 global study, 80 were also randomized in the China extension study for MK-7902-007 (NCT04676412).
Groups:
- Pembrolizumab + Lenvatinib: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily (QD) on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity. As of 30-Jul-2021, participants discontinued lenvatinib and participants who remained on treatment received open-label pembrolizumab only at same dose and schedule.
- Pembrolizumab + Placebo: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule QD on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity. As of 30-Jul-2021, participants discontinued placebo and participants who remained on treatment received open-label pembrolizumab only at same dose and schedule.
Period: Overall Study
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Started | 309 | 314
Treated | 309 | 312
Completed | 0 | 0
Not Completed | 309 | 314
Not completed — Death | 225 | 230
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor Decision | 71 | 72
Not completed — Withdrawal by Subject | 11 | 9

BASELINE CHARACTERISTICS:
Population: All participants randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo | Total
Number analyzed (Participants) | 309 | 314 | 623
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.6) | 65.4 (8.8) | 65.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 90 | 169
  Male | 230 | 224 | 454
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 30 | 62
  Not Hispanic or Latino | 266 | 269 | 535
  Unknown or Not Reported | 11 | 15 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 3 | 10
  Asian | 103 | 104 | 207
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 188 | 193 | 381
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 8 | 10 | 18
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  Participants
    ECOG = 0 | 110 | 108 | 218
    ECOG = 1 | 199 | 206 | 405
Programmed Cell Death Ligand 1 (PD-L1) Status at Baseline [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Randomization of participants in the study was stratified by PD-L1 tumor proportion score (TPS) at baseline (1-49% or ≥ 50%). Higher percentages of PD-L1 TPS staining correspond to higher positivity of PD-L1 on a tumor.
  Participants
    TPS = 1-49% | 172 | 175 | 347
    TPS = ≥ 50% | 137 | 139 | 276
Geographic Region [Count of Participants; unit: Participants] — Randomization of participants in this study was stratified by geographic region of the enrolling site (East Asia or non-East Asia).
  Participants
    East Asia | 103 | 104 | 207
    Non-East Asia | 206 | 210 | 416

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from date of randomization to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Data are from the product-limit (Kaplan-Meier) method for censored data. PFS as assessed by blinded independent central review (BICR) per RECIST 1.1 was presented.
Time Frame: Up to approximately 25 months
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 309 | 314
Months | 6.6 [6.1 to 8.2] | 4.2 [4.1 to 6.2]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Hazards ratio (HR) and 95% confidence interval (CI) were calculated using Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 Status (1% to 49% versus >=50%); Test type: Other; p = 0.00624, Stratified Log Rank; One-sided p-value based on log-rank test stratified by ECOG, region and baseline PD-L1 status; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.64 to 0.95]

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to date of death from any cause. OS was presented.
Time Frame: Up to approximately 25 months
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 309 | 314
Months | 14.1 [11.4 to 19.0] | 16.4 [12.6 to 20.6]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; HR and 95% CI were calculated using Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 Status (1% to 49% versus >=50%); Test type: Other; p = 0.79744, Stratified Log Rank; One-sided p-value based on log-rank test stratified by ECOG, region, and baseline PD-L1 status; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.87 to 1.39]

3. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR as assessed by BICR per RECIST 1.1 is presented.
Time Frame: Up to approximately 25 months
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 309 | 314
Percentage of Participants | 40.5 [34.9 to 46.2] | 27.7 [22.8 to 33.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Percent difference and 95% CI were calculated using Miettinen & Nurminen method stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 Status (1% to 49% versus >=50%); Test type: Other; p = 0.00037, Stratified Miettinen & Nurminen; One-sided p-value for testing. H0: difference in percent = 0 versus H1: difference in percent > 0; Percent Difference = 12.8, 95% CI 2-sided [5.4 to 20.1]

4. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced an AE were reported
Time Frame: Through 90 days post last dose of study treatment (Up to approximately 27 months)
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 309 | 312
Participants | 306 | 294

5. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued study treatment due to an AE were reported.
Time Frame: Through last dose of study treatment (Up to approximately 24 months)
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 309 | 312
Participants | 98 | 41

6. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment (EORTC) Quality of Life Questionnaire-Core30 (QLQ-C30) Combined Global Health Status/Quality of Life (Items 29 & 30) Scale Combined Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall quality of life (QoL) of cancer patients. Participant responses to questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) is computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. Per protocol, the change from baseline in GHS and QoL combined score was presented.
Time Frame: Baseline and Week 21
Population: All randomized participants who have received at least one dose of the study intervention and had at least one EORTC QLQ-C30 assessment data available for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 309 | 308
Score on a scale | -1.48 [-4.09 to 1.13] | 2.42 [-0.24 to 5.08]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — Difference in LS means and 95% CI were calculated using the Constrained longitudinal data analysis (cLDA) model with covariates for treatment by study visit interaction & stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 Status (1% to 49% versus >=50%); p = 0.0262, Constrained longitudinal data analysis; Two-sided p-value based on cLDA model with covariates for treatment by study visit interaction; stratified by ECOG, region & baseline PDL-1; Difference in Least Square (LS) Means = -3.90, 95% CI 2-sided [-7.34 to -0.47]

7. Secondary Outcome: Change From Baseline in Cough (EORTC Quality of Life Questionnaire-Lung Cancer Module 13 [QLQ-LC13] Item 31) Score
Description: The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. Per protocol, the change from baseline in cough (EORTC QLQ-LC13 Item 31) score was presented.
Time Frame: Baseline and Week 21
Population: All randomized participants who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Item 31 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 309 | 307
Score on a scale | -9.53 [-12.94 to -6.13] | -5.04 [-8.51 to -1.57]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — Difference in LS means and 95% CI were calculated using the cLDA model with covariates for treatment by study visit interaction & stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 Status (1% to 49% versus >=50%); p = 0.0461, cLDA model — Two-sided p-value based on cLDA model with covariates for treatment by study visit interaction; stratified by ECOG, region & baseline PDL-1; Difference in LS means = -4.50, 95% CI 2-sided [-8.91 to -0.08]

8. Secondary Outcome: Change From Baseline in Chest Pain (EORTC QLQ-LC13 Item 40) Score
Description: The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. Per protocol, the change from baseline in EORTC QLQ-LC13 chest pain (Item 40) score was presented.
Time Frame: Baseline and Week 21
Population: All randomized participants who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Item 40 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 309 | 307
Score on a scale | -4.64 [-7.45 to -1.84] | -3.55 [-6.42 to -0.68]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.5596, cLDA model; [statistical method as in outcome 6, analysis 1]; Difference in LS means = -1.10, 95% CI 2-sided [-4.78 to 2.59]

9. Secondary Outcome: Change From Baseline in Dyspnea (EORTC QLQ-C30 Item 8) Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to the question: "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. Per protocol, the change from baseline in EORTC QLQ-C30 dyspnea (Item 8) score was presented.
Time Frame: Baseline and Week 21
Population: All randomized participants who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Item 8 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 309 | 308
Score on a scale | -1.35 [-4.75 to 2.04] | -0.47 [-3.94 to 3.00]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.7088, cLDA model; [statistical method as in outcome 6, analysis 1]; Difference in LS means = -0.88, 95% CI 2-sided [-5.49 to 3.74]

10. Secondary Outcome: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. Per protocol, the change from baseline in EORTC QLQ-C30 physical functioning (Items 1-5) combined score was presented.
Time Frame: Baseline and Week 21
Population: All randomized participants who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Items 1-5 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 309 | 308
Score on a scale | -6.73 [-9.35 to -4.10] | -3.72 [-6.40 to -1.04]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.1116, cLDA model; [statistical method as in outcome 6, analysis 1]; Difference in LS means = -3.01, 95% CI 2-sided [-6.71 to 0.70]

11. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-C30 Combined Global Health Status /Quality of Life (Items 29 & 30) Scale Combined Score
Description: EORTC QLQ-C30 is a questionnaire to assess QoL of cancer patients. Participant responses to questions on GHS ("How would you rate your overall health during the past week?") and QoL ("How would you rate your overall QoL during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) was computed by averaging raw scores of the 2 items and applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in GHS-QoL combined score. A longer TTD indicates a better outcome.
Time Frame: Up to approximately 25 months
Population: All randomized participants who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Item 29 and Item 30 assessment data available.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 304 | 297
Months | NA [14.1 to NA] — NA = Median and upper limit of 95%CI was not reached due to insufficient number of participants with an event. | NA [19.3 to NA] — NA = Median and upper limit of 95%CI was not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — HR and 95% CI were calculated using Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 Status (1% to 49% versus >=50%); p = 0.9601, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG, region and baseline PD-L1 status; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.75 to 1.33]

12. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-LC13 Cough (Item 31) Scale Score
Description: EORTC QLQ-LC13 is a lung cancer specific questionnaire. Participant responses to the question: "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0-100. A lower score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in cough (Item 31). A longer TTD indicates a better outcome.
Time Frame: Up to approximately 25 months
Population: All randomized participants who received at least one dose of study treatment and have at least one EORTC-QLQ-LC13 Item assessment data available.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 304 | 294
Months | NA [NA to NA] — NA = Median, lower and upper limit of 95%CI was not reached due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower and upper limit of 95%CI was not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.0079, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG, region and baseline PD-L1 status; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.42 to 0.88]

13. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-LC13 Chest Pain (Item 40) Scale Score
Description: EORTC QLQ-LC13 is a lung cancer specific questionnaire. Participant responses to the question: "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0-100. A lower score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in cough (Item 40). A longer TTD indicates a better outcome.
Time Frame: Up to approximately 25 months
Population: All randomized participants who received at least one dose of study treatment and have at least one EORTC-QLQ-LC13 Item 40 assessment data available.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 304 | 294
Months | NA [NA to NA] — NA = Median, lower and upper limit of 95%CI were not reached due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower and upper limit of 95%CI were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.7457, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG, region and baseline PD-L1 status; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.73 to 1.56]

14. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-C30 Dyspnea (Item 8) Scale Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to the question: "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in dyspnea (Item 8). A longer TTD indicates a better outcome.
Time Frame: Up to approximately 25 months
Population: All randomized participants who received at least one dose of study treatment and have at least one EORTC-QLQ Item 8 assessment data available.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 304 | 297
Months | NA [NA to NA] — NA = Median, lower and upper limit of 95%CI were not reached due to insufficient number of participants with an event. | NA [20.8 to NA] — NA = Median and upper limit of 95%CI were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.8122, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG, region and baseline PD-L1 status; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.75 to 1.44]

15. Secondary Outcome: Time to True Deterioration (TTD) Based on Change From Baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in physical functioning (Items 1 to 5). A longer TTD indicates a better outcome.
Time Frame: Up to approximately 25 months
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 304 | 297
Months | 18.8 [14.1 to NA] — NA = Upper limit of 95%CI could not be reached due to insufficient number of participants with an event. | NA [20.0 to NA] — NA = Median and upper limit of 95%CI could not be reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.1480, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG, region and baseline PD-L1 status; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.92 to 1.67]

16. Secondary Outcome: Time to True Deterioration (TTD) Based on Change From Baseline in the Composite Endpoint of Cough (EORTC QLQ-LC13 Item 31), Chest Pain (EORTC QLQ-LC13 Item 40), or Dyspnea (EORTC QLQ-C30 Item 8)
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients, including a single-item scale score for dyspnea (Item 8; score range:1=Not at All to 4=Very Much). Used in combination with QLQ-C30, the EORTC QLQ-LC13 is a supplemental lung cancer-specific module, including a single-item scale score for cough (Item 31; score range:1=Not at All to 4=Very Much ) and chest pain (Item 40, score range: 1=Not at All to 4=Very Much). The combined score of items 31, 40 and 8 was computed by averaging the raw scores of the items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. The TTD in the composite endpoint of EORTC QLQ-LC13 Item 31, EORTC QLQ-LC13 Item 40, EORTC QLQ-C30 Item 8 scale score was presented, defined as the time to first onset of a ≥10point decrease from baseline in anyone of the three scale items. A longer TTD indicates better outcome.
Time Frame: Up to approximately 25 months
Population: All randomized participants who received at least one dose of study treatment and have at least one had at least one EORTC-QLQ-C30 or EORTC QLQ-LC13 assessment data available.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Months | 5.78 [2.79 to NA] — NA = Upper limit of 95%CI could not be reached due to insufficient number of participants with an event. | NA [3.45 to NA] — NA = Median and upper limit of 95%CI could not be reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 11, analysis 1]; p = 0.4068, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG, region and baseline PD-L1 status; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.70 to 2.46]

ADVERSE EVENTS:
Time Frame: Up to approximately 61 months
Description: All-Cause Mortality includes all randomized participants. Serious and Other adverse events (AEs) includes all randomized participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Groups:
- Lenvatinib + Pembrolizumab: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily (QD) on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity. As of 30-Jul-2021, participants discontinued lenvatinib and participants who remained on treatment received open-label pembrolizumab only at same dose and schedule.
- Placebo + Pembrolizumab: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule QD on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity. As of 30-Jul-2021, participants discontinued placebo and participants who remained on treatment received open-label pembrolizumab only at same dose and schedule.
Arm/Group | Lenvatinib + Pembrolizumab | Placebo + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 229/309 | 232/314
Serious Adverse Events (participants affected / at risk) | 192/309 | 118/312
Other Adverse Events (participants affected / at risk) | 296/309 | 275/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=309) | Placebo + Pembrolizumab (N=312)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 3 (3)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4) | 1 (2)
Colitis ulcerative (Gastrointestinal disorders) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral cavity fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 4 (5) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 5 (5) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1)
Death (General disorders) | 13 (13) | 1 (1)
Fatigue (General disorders) | 5 (5) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Polyserositis (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Strangulated hernia (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 8 (8) | 4 (5)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 2 (3) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 32 (38) | 17 (19)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Amylase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Coagulation time prolonged (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 3 (3) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 4 (4)
Demyelination (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (2)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vancomycin infusion reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=309) | Placebo + Pembrolizumab (N=312)
Anaemia (Blood and lymphatic system disorders) | 57 (84) | 68 (88)
Hyperthyroidism (Endocrine disorders) | 30 (35) | 20 (25)
Hypothyroidism (Endocrine disorders) | 127 (171) | 35 (36)
Abdominal pain (Gastrointestinal disorders) | 27 (33) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 24 (27) | 13 (13)
Constipation (Gastrointestinal disorders) | 37 (42) | 44 (50)
Diarrhoea (Gastrointestinal disorders) | 109 (208) | 39 (62)
Nausea (Gastrointestinal disorders) | 70 (116) | 42 (76)
Stomatitis (Gastrointestinal disorders) | 52 (71) | 12 (12)
Vomiting (Gastrointestinal disorders) | 35 (56) | 17 (26)
Asthenia (General disorders) | 57 (86) | 35 (37)
Chest pain (General disorders) | 23 (26) | 15 (15)
Fatigue (General disorders) | 44 (58) | 37 (40)
Oedema peripheral (General disorders) | 31 (42) | 18 (20)
Pyrexia (General disorders) | 33 (42) | 32 (41)
Pneumonia (Infections and infestations) | 27 (28) | 14 (15)
Urinary tract infection (Infections and infestations) | 25 (39) | 19 (33)
Alanine aminotransferase increased (Investigations) | 60 (79) | 32 (42)
Amylase increased (Investigations) | 30 (45) | 10 (11)
Aspartate aminotransferase increased (Investigations) | 62 (89) | 32 (49)
Blood alkaline phosphatase increased (Investigations) | 35 (47) | 17 (29)
Blood creatinine increased (Investigations) | 23 (27) | 19 (23)
Blood thyroid stimulating hormone increased (Investigations) | 24 (29) | 7 (11)
Lipase increased (Investigations) | 29 (50) | 15 (18)
Platelet count decreased (Investigations) | 32 (46) | 7 (11)
Weight decreased (Investigations) | 83 (98) | 25 (27)
Decreased appetite (Metabolism and nutrition disorders) | 77 (92) | 51 (55)
Hyperglycaemia (Metabolism and nutrition disorders) | 25 (39) | 23 (30)
Hyperkalaemia (Metabolism and nutrition disorders) | 17 (20) | 12 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 34 (39) | 20 (31)
Hypocalcaemia (Metabolism and nutrition disorders) | 24 (31) | 11 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 28 (34) | 23 (28)
Hyponatraemia (Metabolism and nutrition disorders) | 37 (49) | 23 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 (50) | 33 (43)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (28) | 24 (26)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (20) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (23) | 14 (16)
Dizziness (Nervous system disorders) | 19 (25) | 10 (11)
Headache (Nervous system disorders) | 28 (40) | 13 (13)
Insomnia (Psychiatric disorders) | 17 (18) | 13 (13)
Haematuria (Renal and urinary disorders) | 22 (30) | 17 (25)
Proteinuria (Renal and urinary disorders) | 101 (169) | 36 (55)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (38) | 25 (27)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 (36) | 27 (29)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 25 (29) | 27 (49)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 34 (37) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 33 (44) | 29 (33)
Rash (Skin and subcutaneous tissue disorders) | 44 (57) | 33 (37)
Hypertension (Vascular disorders) | 122 (150) | 46 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT03829332/Prot_SAP_001.pdf